CLINICAL TRIAL: NCT05541367
Title: Estrogen Receptor (ER) PET/CT Imaging in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJ-IRB20211128
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; TNBC - Triple-Negative Breast Cancer; Estrogen-receptor-negative Breast Cancer
Keywords: Estrogen receptor; PET/CT; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
18F-Fluoroestradiol (18F-FES) is an estrogen receptor-targeting positron emission tomography tracer with high sensitivity and specificity for the detection of estrogen receptor（ER）-positive tumors . 18F-FES has been used as a predictive biomarker to demonstrate estrogen receptor heterogeneity , to evaluate the pharmacokinetics of estrogen receptor-targeted drugs ， to measure residual estrogen receptors during endocrine therapy and to determine biologically optimal doses of novel estrogen receptor-targeted drugs .This study aimes to explore the efficacy of 18F-FES PET/CT in evaluating the expression levels of ER in primary and metastatic breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women, and up to 70% of breast cancer patients are positive for hormone receptors. Most of them are estrogen receptor (ER) positive, and more than 95% of progesterone receptor (PR) positive tumors are also ER positive. The staging system most commonly used for BC is the American Joint Committee on Cancer TNM system, which is based on seven criteria - tumor extent (T), spread to nearby lymph nodes (N), spread (metastasis) to distant sites (M), cancer grade ( G), estrogen receptor (ER) status, progesterone receptor status (PR) and HER2/neu . Breast cancer is characterized by different pathological features, different responses to treatment, and significant differences in long-term survival among patients . In general, the molecular typing of breast cancer is mainly divided into four types: the first, luminalA type refers to ER, PR positive, HER2 negative, and endocrine therapy can be performed. The second, luminalB type means that ER, PR and HER2 are all positive, endocrine therapy, chemotherapy and targeted therapy can be used, and the therapeutic effect is relatively good. The third type, HER2 overexpression type is HER2 positive, ER and PR are both negative, this type is ineffective for endocrine therapy, and targeted therapy can be used. Fourth, ER, PR and HER2 are all negative , and the treatment effect is the worst. In general, the two subtypes of luminalA and B have higher long-term survival rates. Meanwhile,HER2 overexpression and triple-negative breast cancer have a poor prognosis.

The success of breast cancer treatment depends heavily on tumor estrogen receptor status, which is currently assessed by immunohistochemistry. While immunohistochemistry is well suited to detect primary breast tumors, metastatic foci are less accurate. Estrogen receptor expression changes over time, and inconsistent expression between primary and metastatic tumors has been observed in up to 40% of patients.Studies have shown the potential role of FES-PET/CT in assessing ER status, especially in patients with multiple tumors or that are difficult to biopsy.FES-PET/CT as an imaging technique targeting estrogen receptors may help predict patient response to endocrine therapy. Therefore, FES PET/CT imaging is of great significance for the selection of patients who benefit from endocrine therapy and those who are better through adjuvant chemotherapy .

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Patients with pathologically confirmed breast cancer
* Sign the informed consent form

Exclusion Criteria:

* Pregnant women
* Severe underlying diseases that cannot cooperate with PET examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients should be more than 18 years old,and have been pathologically confirmed breast cancer.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 5 years
  SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: ZHU XIAOHUA, DR, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China